CLINICAL TRIAL: NCT02640521
Title: Pilot Testing an Intervention to Increase Implementation of Evidence-based Guidelines to Achieve Smoking Cessation in Smoking Parents of Inner-city Children With Asthma
Brief Title: Smoking Cessation Peds Asthma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Lincoln Medical and Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-00742
Record Dates: First submitted 2015-12-16; First posted 2015-12-29 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Smoking Cessation; Asthma
MeSH Terms: conditions — Smoking Cessation; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Parents (No Intervention)
- Treatment Parents (Active Comparator): Chart reminders (paper or electronic medical records, depending on clinic wishes) to prompt providers to ask about in home smoking at every medical visit; establishing a New York State Quit line referral system in the pediatric practice; and amending the training curriculum for providers and the patient education materials that are part of a provider toolkit, to focus on the negative impact of second hand smoke (SHS) on their children,and specifically, asthma outcomes.
  Interventions: Behavioral: Chart Reminders & New York State Quit line referral system

INTERVENTIONS:
Behavioral: Chart Reminders & New York State Quit line referral system — Investigators at New York University Medical School, Bellevue and Lincoln Hospital will work closely to (1) develop chart reminders appropriate for each of their clinics (2) to prompt providers to ask about in home smoking at every medical visit and (3) to establish a New York Quit line referral system in the pediatric practice, including clearly defined roles and responsibilities for each step. The New York State Quit line service includes proactive telephone calls with mailings of self-help material, free nicotine replacement therapy for those who qualify, and referrals to local treatment programs, ensuring that health literacy levels of materials is maximized, amending the training curriculum for providers as necessary, and modifying patient education materials that are part of the provider tool kit to focus on the negative impact of secondhand smoke.
  Arms: Treatment Parents

SUMMARY:
The overall goal of this study is to adapt and preliminarily validate an intervention based on evidence based approaches to assist smoking parents and other family members of inner-city children ages 4 to 12 with asthma to stop smoking.This study aims (1) to adapt existing guideline-based materials used in adult medicine to create a system- and provider-level intervention for pediatrics and (2) to evaluate feasibility and acceptability of (a) procedures to recruit inner-city, ethnic minority parents and (b) intervention procedures, and to estimate intervention effects.

DETAILED DESCRIPTION:
Investigators will adapt guideline-based interventions used in adult medicine. The intervention consists of two system-level interventions (chart reminders to prompt providers to ask about in-home smoking and a State Quit-line referral system), and a provider-level intervention (training in the PHS Guidelines, in motivational interviewing, and on how to use the system-level intervention). Investigators will implement the study in the Bellevue Pediatric Asthma Clinic and the pediatric clinic at Lincoln Hospital using a two group (pre intervention control group / post-intervention treatment group) pilot study to test the feasibility and preliminary effects of a multi-level (i.e., system and provider) intervention. The primary outcome is provider adherence to tobacco use treatment guidelines, which will be assessed by conducting parent exit interviews with 200 smoking parents (100 pre-intervention [control group] and 100 post-intervention [treatment group]). Preliminary intervention outcomes will be collected through the parent exit interviews (i.e., baseline) and 2-month post-baseline interviews with the control and treatment parents. Providers will also be interviewed regarding their satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Parents of a child between the ages of 4 and 12 with uncontrolled asthma, brought to one of the clinics for an asthma-related visit
* uncontrolled asthma as meeting the criteria for "not well-controlled" or "very poorly controlled" asthma: (a) score of 19 or lower on the validated Asthma Control Test (ACT)45 OR (b) any of the following in the prior 12 months: (1) 2+ courses of oral steroids; (ii) 2+ Emergency Department (ED) visits for asthma; and (iii) 1+ hospitalization for asthma.
* The parents must speak English or Spanish, and have the capacity to provide consent.

Exclusion Criteria:

* Beyond these eligibility criteria, no exclusions will be made based on sex, ethnicity, or race of the child or parent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of pre-intervention patients that adhere to to Public Health Service (PHS) Guidelines from Providers | 2-Month Follow Up

SECONDARY OUTCOMES:
Change in score of Asthma Control Test | 2- Month Follow-Up
Frequency of medication use in the prior 2 months | 2- Month Follow-Up
Frequency of unscheduled clinic visits | 2- Month Follow-Up
Frequency of Emergency Department visits for asthma in prior 2 months | 2- Month Follow-Up
Frequency of hospitalizations for asthma in prior 2 month | 2- Month Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marie Bruzzese, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States